CLINICAL TRIAL: NCT07099261
Title: A Comparative Clinical Study to Evaluate Crowns Designed by Artificial Intelligence Versus a Crowns Designed Traditional Design Software
Brief Title: A Comparative Clinical Study to Evaluate Crowns Designed by Artificial Intelligence Versus Crowns Designed Traditional Design Software
Acronym: AI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Tishreen U ـProsthodontics
Record Dates: First submitted 2025-07-20; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Dental Crown
Keywords: Crowns; Crowns Designed by Artificial Intelligence; Artificial intelligence(AI); CAD; CAD\CAM; computer-aided design and computer-aided manufacturing; prosthesis
MeSH Terms: interventions — Crowns

STUDY DESIGN:
Intervention Model Description: self controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crowns designed with AI powered dentibird (Experimental): 10 Crowns designed with AI powered dentbird
  Interventions: Other: Crowns
- Crowns designed with AI powered Exocad (Experimental): 10 Crowns designed with AI powered Exocad
  Interventions: Other: Crowns
- Crowns designed with conventional Exocad (Sham Comparator): 10 Crowns designed with conventional Exocad (computer aided experienced)
  Interventions: Other: Crowns

INTERVENTIONS:
Other: Crowns — 1. Tooth Preparation: Prepare the teeth to receive a zirconia crown.
  2. Impression Taking: Obtain impressions using silicone.
  3. Digital Conversion: Convert impressions into a digital model using a laboratory scanner.
  4. Design Submission: Send the digital model to selected crown design program.
  5. Crown Fabrication: crowns designed will be produced from PMMA using a milling unit.
  6. Clinical Evaluation: Conduct a clinical assessment of the crowns
  7. the best crown design will be milled from zirconia and delivered
  Evaluation of Crowns designed by following metrics:
  1. Marginal fit
  2. proximal contact
  3. Occlusion
  Other Names: dental crowns

SUMMARY:
This clinical research aims to Evaluate Crowns Designed by Artificial Intelligence Versus Crowns Designed by Traditional Design Software

The research will be conducted on a sample of patients with an indication for crowning of the first lower molar. Ten dental crowns will be prepared.

After obtaining written consent from patients who meet the inclusion and exclusion criteria, 10 dental crowns will be prepared. Measurements will be taken using silicone impressions and then converted into digital format.

The digital impression will be sent to the selected dental restoration design software used in the study. The same parameters will be adjusted in all software programs for each crown.

After the design is completed, the designs will be sent to the milling unit. For each case, three crowns will be designed and milled from polymethyl methacrylate (PMMA).

The crown will be clinically examined and evaluated according to specific criteria. Marginal fit, proximal contact quality, and occlusion will be assessed.

The best crown will be milled from zirconia and delivered to the patient.

DETAILED DESCRIPTION:
Recent advancements in artificial intelligence (AI) have revolutionized various fields, including dentistry, where AI systems are being promoted to reduce design time for dental restorations. However, it remains unclear whether this increased speed compromises critical factors such as marginal fit accuracy, occlusion, and contact points-elements crucial for the success of dental prosthetics. The existing scientific evidence regarding the efficiency of AI-supported dental design systems is limited. A review of the literature revealed only one clinical study addressing this aspect, highlighting the urgent need for further comparative research.

This clinical research aims to Evaluate Crowns Designed by two Artificial Intelligence computer-aided AIـCAD Versus Crowns Designed by Traditional Design Software One Traditional CAD by assessing the following metrics:

1. Marginal fit accuracy
2. Quality of contact points
3. Occlusion

Importance of the Research

Given the scarcity of studies focusing on AI-based crown design systems clinically, this research will assist dental clinics and laboratories in making informed decisions regarding the adoption of AI technologies versus continuing with traditional methodologies.

Study Design

self controlled clinical trial

Clinical Procedures

1. Tooth Preparation: Prepare the teeth to receive a zirconia crown.
2. Impression Taking: Obtain impressions using silicone.
3. Digital Conversion: Convert impressions into a digital model using a laboratory scanner.
4. Designing : Send the digital model to selected crown design programs (both AI-driven and traditional).
5. Crown Fabrication: After design approval, crowns will be produced from PMMA using a milling unit.
6. Clinical Evaluation: Conduct a clinical assessment of the crowns. Evaluation Metrics

Marginal Fit Accuracy

Measurement clinically using a probe. Comparison with silicone replica technique or Analysis through 3D modeling software (X control GEOM).

Contact Points Quality

Measure the force required to pull a dental floss between teeth.

Occlusion Assessment

Utilize 100-micron and 12-micron articulating paper and Shimstock to evaluate occlusal contact points.

Data will be analyzed using appropriate statistical methods to compare the outcomes between AI-driven designs and traditional methods, ensuring robust conclusions regarding their efficacy.

The results of this study are anticipated to provide valuable insights into the reliability and quality of AI-based crown design systems compared to traditional methods, guiding dental practices in their decision-making processes regarding technology adoption.

This proposal serves as a foundation for conducting a thorough investigation into the effectiveness of AI in dental crown design, addressing a critical gap in current research and practice

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years requiring a crown for a lower first molar
* Good oral and gingival health
* adjacent teeth in good condition
* Natural opposing teeth
* Willingness to participate and sign informed consent

Exclusion Criteria:

* Abnormal occlusal habits such as bruxism
* Active periodontal diseases
* Allergy to crown materials (e.g., polymethyl methacrylate, PMMA)
* Poor oral hygiene

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Marginal Fit | immediately after delivering the crown
  Evaluation is conducted by 2 dentists to determine whether the restoration is clinically acceptable or unacceptable using an explorer
  or The silicone replica technique (Silicone Replica Technique) is used to evaluate the marginal fit of crowns using silicone material
  or Evaluation is conducted using Geomagic X
Clinical evaluation of proximal contact points | immediately after delivering the crown
  To evaluate the interproximal contact points of the crown clinically using waxed dental floss: if the floss passes with slight resistance, the contact points are considered acceptable if the floss passes without resistance, the contact points are considered unacceptable if the floss hard to pass or tearing, the contact points are considered Tight Contact
clinical evaluation of the occlusion | immediately after delivering the crown
  Clinical Evaluation of Occlusion Using Articulating Paper Excellent (both 100- and 12-mm articulating paper imprints exist on the crown and adjacent teeth) nice occlusal contact distribution Good (only 100-mm articulating paper imprints exist on adjacent teeth) Individual occlusal contact points missing or deviated but occlusal contacts on main supporting cusp Satisfactory crown too high, thus supra occlusion No occlusal contacts on supporting cusps but contacts present on other parts of occlusal surface
  Unsatisfactory No occlusal contact points on crown(infra occlusion)

CONTACTS AND LOCATIONS:
Overall Officials: Zeyad Handhal, master's student, Principal Investigator — Tishreen University; Rima Saker, Assistant professor, Study Chair — Tishreen University

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet

REFERENCES:
- See also: Evaluation of the accuracy, occlusal contact and clinical applications of zirconia crowns using artificial intelligence design versus human design — https://doi.org/10.1016/j.jds.2025.03.016
- See also: Impact of different CAD software programs on marginal and internal fit of provisional crowns: An in vitro study — https://doi.org/10.1016/j.heliyon.2024.e24205
- See also: Time efficiency, occlusal morphology, and internal fit of anatomic contour crowns designed by dental software powered by generative adversarial network: A comparative study — https://doi.org/10.1016/j.jdent.2023.104739
- See also: Verification of the accuracy and design time of crowns designed with artificial intelligence — https://doi.org/10.4047/jap.2025.17.1.1